CLINICAL TRIAL: NCT00820248
Title: A Phase III Study of Standard Fractionation Radiotherapy With Concurrent High-Dose Cisplatin Versus Accelerated Fractionation Radiotherapy With Panitumumab in Patients With Locally Advanced Stage III and IV Squamous Cell Carcinoma of the Head and Neck
Brief Title: Radiation + Cisplatin or Panitumumab in Locally Advanced Stage III or Stage IV Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HN6; CAN-NCIC-HN6 (Registry Identifier: NCI US - Physician Data Query); CDR0000630159 (Other: PDQ)
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2020-04

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the oropharynx; stage III verrucous carcinoma of the oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV verrucous carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Panitumumab; Cisplatin; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Active Comparator): Patients undergo standard fractionation radiotherapy (IMRT or 3D CRT) once daily, 5 days a week, for 7 weeks. Patients receive cisplatin IV over 1 hour on days 1, 22, and 43 of radiotherapy.
  Interventions: Drug: cisplatin; Radiation: 3-dimensional conformal radiation therapy; Radiation: intensity-modulated radiation therapy
- Arm II (Experimental): Patients undergo accelerated fractionation radiotherapy (IMRT or 3D CRT) once or twice daily, 5 days a week, for 6 weeks. Patients receive panitumumab IV over 30-90 minutes 1 week prior to and on days 15 and 36 of radiotherapy.
  Interventions: Biological: panitumumab; Radiation: 3-dimensional conformal radiation therapy; Radiation: accelerated radiation therapy; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Biological: panitumumab — Given IV
  Arms: Arm II
Drug: cisplatin — Given IV
  Arms: Arm I
Radiation: 3-dimensional conformal radiation therapy — Patients undergo radiotherapy
Radiation: accelerated radiation therapy — Patients undergo accelerated fractionation radiotherapy
  Arms: Arm II
Radiation: intensity-modulated radiation therapy — Patients undergo radiotherapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy in higher doses over a shorter period of time may kill more tumor cells and have fewer side effects. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as panitumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether giving standard radiation therapy together with high-dose cisplatin is more effective than giving higher-dose radiation therapy together with panitumumab in treating patients with locally advanced head and neck cancer.

PURPOSE: This randomized phase III trial is comparing two radiation therapy regimens to see how well they work when given together with cisplatin or panitumumab in treating patients with locally advanced stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the progression-free survival (PFS) of patients with locally advanced squamous cell carcinoma of the head and neck treated with standard fractionation radiotherapy and high-dose cisplatin vs accelerated fractionation radiotherapy and panitumumab.

Secondary

* To compare overall survival of patients treated with these regimens.
* To compare local and regional PFS of patients treated with these regimens.
* To compare distant metastasis in patients treated with these regimens.
* To compare adverse events, including late radiotherapy-related adverse events in patients treated with these regimens.
* To compare quality of life (QOL) of patients treated with these regimens.
* To compare swallowing-related QOL of patients treated with these regimens.
* To compare economic evaluation (cost effectiveness analysis and cost utility), including both healthcare utilization and indirect costs.

OUTLINE: This is a multicenter study. Patients are stratified according to T category (T1-3 vs T4), nodal status (N0-1 vs N2 vs N3), radiotherapy delivery modality (intensity-modulated [IMRT] vs 3-D conformal [3D CRT]), anatomic location (hypopharynx vs oral cavity vs oropharynx vs larynx), and participation in the optional swallowing impairment substudy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo standard fractionation radiotherapy (IMRT or 3D CRT) once daily, 5 days a week, for 7 weeks. Patients receive cisplatin IV over 1 hour on days 1, 22, and 43 of radiotherapy.
* Arm II: Patients undergo accelerated fractionation radiotherapy (IMRT or 3D CRT) once or twice daily, 5 days a week, for 6 weeks. Patients receive panitumumab IV over 30-90 minutes 1 week prior to and on days 15 and 36 of radiotherapy.

Treatment in both arms continues in the absence of disease progression or unacceptable toxicity.

Quality of life (QOL) (FACT-H&N), swallowing-related QOL (MDADI, SWAL-QOL), swallowing function (FOIS), and economic evaluations (Lost Productivity questionnaire) are assessed periodically during the study.

After completion of study treatment, patients are followed periodically for at least 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically and/or cytologically confirmed (primary lesion or regional lymph nodes) squamous cell carcinoma of the oral cavity, oropharynx, larynx, or hypopharynx

  * Locally advanced disease, defined by any of the following criteria:

    * Any T, N+, M0
    * T3-4, N0, M0
* No current history of unknown primary squamous cell carcinoma of the head and neck, primary nasopharyngeal, paranasal, or salivary gland tumors of the head and neck

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Absolute granulocyte count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST or ALT ≤ 3 times ULN
* Creatinine clearance > 50 mL/min
* Magnesium > 0.5 mmol/L
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study treatment
* Must be accessible for treatment and follow-up
* Able (sufficiently fluent) and willing to complete the quality of life (QOL) and swallowing QOL questionnaires in either English or French
* Must be assessed by a radiation oncologist and medical oncologist and deemed suitable for study participation
* No other malignancies within the past 5 years, except adequately treated nonmelanoma skin cancer, curatively treated in-situ cancer of the cervix, or other curatively treated solid tumors
* No history of allergic or hypersensitivity reactions to any of the study drugs or their excipients
* No prior or concurrent interstitial lung disease (e.g., pneumonitis or pulmonary fibrosis) on baseline CT scan
* No peripheral neuropathy ≥ grade 2 (CTCAE v3.0)
* No hearing loss/tinnitus ≥ grade 3 (CTCAE v3.0)
* No thromboembolic event within the past 12 months despite being treated with anticoagulation drugs

  * Prior thromboembolic event > 12 months allowed provided patient is stable on anticoagulation or on preventative anticoagulation
* None of the following allowed:

  * Myocardial infarction within the past 12 months
  * Uncontrolled severe congestive heart failure
  * Unstable angina
  * Active cardiomyopathy
  * Unstable ventricular arrhythmia
  * Uncontrolled hypertension
  * Uncontrolled psychiatric disorder
  * Active serious infection
  * Active peptic ulcer disease
  * Any other medical condition that might interfere with protocol therapy delivery

PRIOR CONCURRENT THERAPY:

* No prior surgical treatment except diagnostic biopsy for this disease
* No prior induction chemotherapy for this disease
* No prior radiation to the head and neck region that would result in overlap of fields for this study
* No prior cisplatin or carboplatin chemotherapy
* No prior targeted anti-EGFR therapy of any kind
* At least 30 days since any prior investigational agent
* No concurrent granulocytic growth factors (e.g., filgrastim [G-CSF]) during radiotherapy
* No concurrent erythropoietic growth factors, pilocarpine, amifostine, other anticancer therapy (e.g., cytotoxic agents, biological response modifiers, immunotherapy, or hormonal therapy), or other investigational drug therapy
* The following radiological investigations must be done within 8 weeks of randomization:

  * MRI or CT of the head and neck
  * CT chest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2008-12-30 (Actual); Primary Completion 2015-05-16 (Actual); Study Completion 2017-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lillian L. Siu, MD, FRCPC, Principal Investigator — Princess Margaret Hospital, Canada; John Waldron, MD, Study Chair — Princess Margaret Hospital, Canada
Locations (19):
- Canada (19):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Northeast Cancer Center Health Sciences, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ringash J, Waldron JN, Siu LL, Martino R, Winquist E, Wright JR, Nabid A, Hay JH, Hammond A, Sultanem K, Hotte S, Leong C, El-Gayed AA, Naz F, Ramchandar K, Owen TE, Montenegro A, O'Sullivan B, Chen BE, Parulekar WR. Quality of life and swallowing with standard chemoradiotherapy versus accelerated radiotherapy and panitumumab in locoregionally advanced carcinoma of the head and neck: A phase III randomised trial from the Canadian Cancer Trials Group (HN.6). Eur J Cancer. 2017 Feb;72:192-199. doi: 10.1016/j.ejca.2016.11.008. Epub 2016 Dec 29. PMID 28040660
- [Result] Siu LL, Waldron JN, Chen BE, Winquist E, Wright JR, Nabid A, Hay JH, Ringash J, Liu G, Johnson A, Shenouda G, Chasen M, Pearce A, Butler JB, Breen S, Chen EX, FitzGerald TJ, Childs TJ, Montenegro A, O'Sullivan B, Parulekar WR. Effect of Standard Radiotherapy With Cisplatin vs Accelerated Radiotherapy With Panitumumab in Locoregionally Advanced Squamous Cell Head and Neck Carcinoma: A Randomized Clinical Trial. JAMA Oncol. 2017 Feb 1;3(2):220-226. doi: 10.1001/jamaoncol.2016.4510. PMID 27930762
- [Derived] Cuffe S, Hon H, Tobros K, Espin-Garcia O, Brhane Y, Harland L, Fadhel E, Eng L, LaDelfa A, Waldron J, Siu LL, Chen BE, Xu W, Simmons C, Kassam Z, Montenegro A, Parulekar WR, Liu G. Cancer patients' acceptability of incorporating an epidemiology questionnaire within a clinical trial. Clin Trials. 2015 Jun;12(3):237-45. doi: 10.1177/1740774514568689. Epub 2015 Jan 29. PMID 25633805

RESULTS

PARTICIPANT FLOW:
Groups:
- Cisplatin: Patients undergo standard fractionation radiotherapy (IMRT or 3D CRT) once daily, 5 days a week, for 7 weeks. Patients receive cisplatin IV over 1 hour on days 1, 22, and 43 of radiotherapy.
  cisplatin: Given IV
  3-dimensional conformal radiation therapy: Patients undergo radiotherapy
  intensity-modulated radiation therapy: Patients undergo radiotherapy
- Panitumumab: Patients undergo accelerated fractionation radiotherapy (IMRT or 3D CRT) once or twice daily, 5 days a week, for 6 weeks. Patients receive panitumumab IV over 30-90 minutes 1 week prior to and on days 15 and 36 of radiotherapy.
  panitumumab: Given IV
  3-dimensional conformal radiation therapy: Patients undergo radiotherapy
  accelerated radiation therapy: Patients undergo accelerated fractionation radiotherapy
  intensity-modulated radiation therapy: Patients undergo radiotherapy
Period: Overall Study
Arm/Group | Cisplatin | Panitumumab
Started | 160 | 160
Received Protocol Treatment (Only treated patients were evaluated for adverse event.) | 156 | 159
Completed | 156 | 159
Not Completed | 4 | 1
Not completed — No treated | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cisplatin | Panitumumab | Total
Number analyzed (Participants) | 160 | 160 | 320
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.68 (7.50) | 56.40 (7.43) | 56.54 (7.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 134 | 134 | 268
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 7 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 158 | 150 | 308
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
ECOG Performance Status [Count of Participants; unit: Participants] — Performance Status:
  0: Fully active, able to carry on all pre-disease performance without restriction
  1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    0 | 111 | 115 | 226
    1 | 49 | 45 | 94
Anatomic Location [Count of Participants; unit: Participants]
  Oral Cavity | 2 | 5 | 7
  Oropharynx | 132 | 127 | 259
  Larynx | 18 | 17 | 35
  Hypopharynx | 8 | 11 | 19
Smoking [Count of Participants; unit: Participants]
  No | 47 | 44 | 91
  Yes | 113 | 116 | 229

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Rate
Description: The progression event is defined by first event of the following,
  Local-regional progression or recurrence Distant metastasis Non-protocol RT, chemotherapy, or biologic therapy without documentation of the site of failure Surgery of primary site with tumour present/unknown Neck dissection with tumour present/unknown, > 15 weeks from end of RT Death due to study cancer or from unknown causes or any other reason
  Number of patients with and without progression event will be reported.
Time Frame: 6.2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cisplatin | Panitumumab
Number analyzed (Participants) | 160 | 160
Participants
  PFS event | 50 | 43
  no PFS event | 110 | 117
Statistical Analysis 1: Comparison: Cisplatin vs Panitumumab; The log rank test stratified by the stratification factors at randomization was used to compare the difference in PFS between two treatment arms; Test type: Superiority; p = 0.83, Regression, Cox; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.60 to 1.50] — Hazard ratio of panitumumab vs cisplatin

2. Secondary Outcome: Overall Survival Rate
Description: Overall survival is defined as the time interval between the date of randomization to date of death from any cause (calculated in months). Otherwise, survival is censored at the last date that the patient is known to be alive.
  Number of death and alive patients will be reported.
Time Frame: 6.2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cisplatin | Panitumumab
Number analyzed (Participants) | 160 | 160
Participants
  Death | 43 | 32
  Alive | 117 | 128
Statistical Analysis 1: Comparison: Cisplatin vs Panitumumab; Test type: Superiority; p = 0.66, Log Rank; Cox Proportional Hazard = 0.89, 95% CI 2-sided [0.54 to 1.48] — hazard ratio for panitumumab vs cisplatin

ADVERSE EVENTS:
Time Frame: 6.2 years
Description: Adverse events were collected on patients who have received the protocol treatment, which were 156 patients in Cisplatin arm and 159 patients in Panitumumab arm, as reported in the Participant Flow.
Arm/Group | Cisplatin | Panitumumab
All-Cause Mortality (participants affected / at risk) | 43/160 | 32/160
Serious Adverse Events (participants affected / at risk) | 0/156 | 0/159
Other Adverse Events (participants affected / at risk) | 156/156 | 159/159
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin (N=156) | Panitumumab (N=159)
Hearing (monitoring program) (Ear and labyrinth disorders) | 25 | 5
Hearing (without monitoring program) (Ear and labyrinth disorders) | 50 | 20
Pain External ear (Ear and labyrinth disorders) | 2 | 8
Pain Middle ear (Ear and labyrinth disorders) | 24 | 29
Tinnitus (Ear and labyrinth disorders) | 98 | 18
Hypothyroidism (Endocrine disorders) | 21 | 22
Dry eye (Eye disorders) | 0 | 10
Chelitis (Gastrointestinal disorders) | 1 | 10
Constipation (Gastrointestinal disorders) | 123 | 113
Diarrhea (Gastrointestinal disorders) | 29 | 40
Dry mouth (Gastrointestinal disorders) | 141 | 146
Dysphagia (Gastrointestinal disorders) | 144 | 150
GI - Other (Gastrointestinal disorders) | 13 | 16
Heartburn (Gastrointestinal disorders) | 36 | 48
Mucositis (clinical exam) Oral cavity (Gastrointestinal disorders) | 120 | 120
Mucositis (functional/symptomatic) Oral cavity (Gastrointestinal disorders) | 51 | 55
Nausea (Gastrointestinal disorders) | 136 | 94
Pain Abdomen NOS (Gastrointestinal disorders) | 11 | 12
Pain Oral cavity (Gastrointestinal disorders) | 32 | 45
Salivary gland changes (Gastrointestinal disorders) | 54 | 67
Teeth (Gastrointestinal disorders) | 8 | 6
Vomiting (Gastrointestinal disorders) | 87 | 63
Edema: head and neck (General disorders) | 38 | 67
Edema: limb (General disorders) | 8 | 6
Fatigue (General disorders) | 124 | 123
Fever (General disorders) | 18 | 17
Pain - Other (General disorders) | 26 | 29
Rigors/chills (General disorders) | 4 | 22
Infection - Other (Infections and infestations) | 44 | 39
Infection with normal ANC Catheter-related (Infections and infestations) | 10 | 9
Dermatitis Chemoradiation (Injury, poisoning and procedural complications) | 64 | 80
Dermatitis Radiation (Injury, poisoning and procedural complications) | 94 | 72
Creatinine (Investigations) | 17 | 0
Lymphopenia (Investigations) | 32 | 34
Weight loss (Investigations) | 136 | 127
Anorexia (Metabolism and nutrition disorders) | 74 | 69
Dehydration (Metabolism and nutrition disorders) | 45 | 38
Fibrosis-deep connective tissue (Musculoskeletal and connective tissue disorders) | 9 | 17
Muscle weakness Whole body/generalized (Musculoskeletal and connective tissue disorders) | 6 | 11
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 7 | 9
Pain Back (Musculoskeletal and connective tissue disorders) | 8 | 11
Pain Bone (Musculoskeletal and connective tissue disorders) | 7 | 9
Pain Extremity-limb (Musculoskeletal and connective tissue disorders) | 8 | 2
Pain Joint (Musculoskeletal and connective tissue disorders) | 8 | 10
Pain Neck (Musculoskeletal and connective tissue disorders) | 20 | 29
Trismus (Musculoskeletal and connective tissue disorders) | 20 | 23
Pain Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 25 | 17
Dizziness (Nervous system disorders) | 19 | 10
Neuropathy-motor (Nervous system disorders) | 5 | 8
Neuropathy-sensory (Nervous system disorders) | 61 | 24
Pain Head/headache (Nervous system disorders) | 33 | 34
Taste alteration (Nervous system disorders) | 142 | 139
Insomnia (Psychiatric disorders) | 50 | 46
Mood alteration Anxiety (Psychiatric disorders) | 22 | 32
Mood alteration Depression (Psychiatric disorders) | 12 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 38
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 | 16
Edema, larynx (Respiratory, thoracic and mediastinal disorders) | 29 | 32
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 26 | 4
Mucositis (clinical exam) Pharynx (Respiratory, thoracic and mediastinal disorders) | 52 | 53
Pain Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 81 | 86
Voice changes (Respiratory, thoracic and mediastinal disorders) | 76 | 74
Acne (Skin and subcutaneous tissue disorders) | 1 | 147
Alopecia (Skin and subcutaneous tissue disorders) | 53 | 50
Dermatology - Other (Skin and subcutaneous tissue disorders) | 7 | 35
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 59
Hand-foot (Skin and subcutaneous tissue disorders) | 1 | 25
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 21 | 33
Hypopigmentation (Skin and subcutaneous tissue disorders) | 6 | 11
Induration (Skin and subcutaneous tissue disorders) | 4 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 18
Rash (Skin and subcutaneous tissue disorders) | 15 | 12
Sweating (Skin and subcutaneous tissue disorders) | 2 | 10
Telangiectasia (Skin and subcutaneous tissue disorders) | 12 | 10
Hypertension (Vascular disorders) | 14 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No